CLINICAL TRIAL: NCT00060788
Title: Intergenerational Transmission of Antisocial Behavior
Brief Title: Antisocial Behavior: Passing From Parent to Child to Grandchild
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: 1R01HD42259-1; 1R01HD042259 (NIH)
Record Dates: First submitted 2003-05-13; First posted 2003-05-14 (Estimated); Last update posted 2006-03-07 (Estimated); Status verified 2006-03

CONDITIONS: Dyssocial Behavior; Antisocial Personality Disorder
Keywords: Antisocial behavior; Mauritius Child Health Project; Intergenerational transmission
MeSH Terms: conditions — Antisocial Personality Disorder

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Antisocial behavior often occurs in different generations within the same family. However, it is not known what factors contribute to this passing of antisocial behavior from parent to child to grandchild. This study is part of a project evaluating antisocial behavior in families; it focuses on the passage of such behavior from one generation to the next.

DETAILED DESCRIPTION:
While it is well-known that antisocial behavior runs in families, little is known about the specific mechanisms by which it is transmitted from one generation to the next. This prospective study will examine biological influences on transgenerational continuity and change, and how biology interacts with social factors in modulating the transmission of antisocial behavior. The study is unique in that it includes both mothers and fathers, focuses on early mechanisms, and addresses female as well as male antisocial behavior.

This study is part of the continuing Mauritius Child Health Project. The project began by testing 1,795 children age 3 years old on psychophysiological, behavioral, nutritional, and cognitive measures. Both male and female children were tested. Their parents were also assessed for psychosocial influences. One hundred children then participated in a nutritional, exercise, and educational enrichment intervention from ages 3 to 5 years old. The intervention has been shown to increase physiological arousal and attention at age 11 years and to reduce conduct disorder at age 17 years.

These 3-year-old children are now 30-year-old adults. This study will retest these adults on psychophysiological, psychosocial, cognitive, behavioral, parenting, and antisocial behavior measures. Their previously untested spouses will also be assessed. Finally, many of these adults now have 3-year-old children of their own; these children will be evaluated as well. Measures of life stress, daily hassles, family conflict, mental illness, and criminal behavior will be assessed. Data from the enrichment cohort will be evaluated to determine if the intervention disrupted the intergenerational transmission of antisocial behavior from the second to third generations.

ELIGIBILITY:
Inclusion Criteria:

* Child of a participant tested in previous Mauritius Child Health Project studies

Ages: 36 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 663
Dates: Start 2001-09; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Raine, Principal Investigator — University of Southern California
Locations (1):
- Joint Child Health Project, Quatre Bornes, Mauritius